CLINICAL TRIAL: NCT00265967
Title: Missed Dose Effect of Irbesartan in Hypertensive Patients and Cardiovascular Risk Profile Monitoring Under Irbesartan Treatment
Brief Title: Irbesartan in Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_9917
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

ARMS (1):
- 1 (Experimental): Irbesartan
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: Irbesartan — Irbesartan 150-300 mg/d for 8 weeks

SUMMARY:
Study objectives:

* To demonstrate the effect of irbesartan on the regulation of diastolic blood pressure, in case of missing one dose after a period of administration for 6 to 8 weeks
* To evaluate the safety of irbesartan

ELIGIBILITY:
Inclusion Criteria:

* Having an average value of ≥ 95 mmHg and ≤ 109 mmHg in diastolic blood pressure measurement or an average diastolic blood pressure value of ≥ 85 mmHg in 24-hours arterial blood pressure measurement,
* Received no treatment within the last 3 months.

Exclusion Criteria:

* Premenopausal women having at least one of the following conditions,

  * Not surgically sterile,
  * Are nursing,
  * Having childbearing potential and not using a reasonable contraception method or not thinking to continue the method throughout the study. Reasonable contraception methods are: intrauterine device, oral or implantable or injectable contraception methods. No methods other than these are accepted.
* Patients routinely sleeping within the day since she/he works at nightshift and whose working hours continue in a time shift from midnight to 04:00 A.M.
* Patients with average systolic blood pressure = 180 mmHg in sitting position or average diastolic blood pressure is ≥110 mmHg in sitting position at baseline visit
* Having known or suspected secondary hypertension
* Having renal and/or hepatic failure together with the following laboratory criteria:

  * Having elevated values of SGPT (ALT) or SGOT (ALT) (at least twice the upper limit of normal range)
  * Having serum creatinine levels of > 2.3 mg/dL (or > 203 μmol/L)
* With bilateral renal artery stenosis or single kidney and unilateral renal artery stenosis or those in post-renal transplantation or with single kidney,
* Having symptomatic sodium insufficiency, hypokalemia or hyperkalemia,
* With volume deficiency,
* With primary hyperaldosteronism,
* With biliary obstructive disorders,
* Having congestive heart failure (New York Heart Association (NYHA)-functional class CHF III-IV),
* With unstable angina pectoris occurring within 3 months before he or she signed the informed consent.
* With stroke occurring within 6 months before he or she signed the informed consent,
* With myocardial infarction or having cardiac surgery within three months before he or she signed the informed consent,
* Underwent PTCA (percutaneous transluminal coronary revascularization) within three months before he or she signed the informed consent,
* Having continuous tachycardia, atrial fibrillation, atrial flutter or other clinical arrythmias defined by the investigator
* With hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically related aortic or mitral valve stenosis,
* With insulin-dependant diabetes mellitus whose blood sugar regulation could not be controlled within the last 3 months after a HbA1C measurement in which it is equal to 10%.
* With a history of drug or alcohol addiction within the last 6 months before she or he signed the informed consent,
* Receiving a drug other than those defined in protocol for blood pressure regulation,
* Who have been participated in any investigational study within the prior month before she or he signed the informed consent
* With a known hypersensitivity against any drug which will be used.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-09; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Changes in 24 hours mean ambulatory blood pressure on the missing dose day. Frequency, severity, seriousness of adverse events emerging during the treatment , and their relation with the study drug. | at the end of 6th months to 8th

SECONDARY OUTCOMES:
Diastolic blood pressure measurements recorded in patients' diaries, and during visits. | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)